CLINICAL TRIAL: NCT02305901
Title: The Effect of Multiple Doses of BI 187004 on the Single-dose Pharmacokinetics of Repaglinide and Bupropion Following Oral Administration in Healthy Male Subjects (an Open-label, One-sequence Trial)
Brief Title: The Effect of Multiple Doses of BI 187004 on the Single-dose Pharmacokinetics of Repaglinide and Bupropion in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1307.20; 2013-005030-38 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
MeSH Terms: interventions — repaglinide

ARMS (1):
- Repaglinide + Bupropion + BI 187004 (Experimental): repaglinide tablets and bupropion tablets with and without concomitant administration of BI 187004
  Interventions: Drug: repaglinide; Drug: BI 187004 tablet; Drug: bupropion extended release tablet

INTERVENTIONS:
Drug: repaglinide — single dose on day 1 of visits 2 and 3
Drug: BI 187004 tablet — multiple doses on days 8-13 of visit 2 and days 1-7 of visit 3
Drug: bupropion extended release tablet — single dose on day 3 of visits 2 and 3

SUMMARY:
To assess the influence of BI 187004 on pharmacokinetics of CYP2C8 and CYP2B6 probe drugs repaglinide and bupropion as a means of predicting drug-drug interactions.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
2. Age of 18 to 55 years (incl.)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders

Further exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of repaglinide in plasma over the time interval from 0 to the last quantifiable data point | up to 48 h post dose
Maximum measured concentration of repaglinide in plasma | up to 48 h post dose
Area under the concentration-time curve of total bupropion in plasma over the time interval from 0 to the last quantifiable data point | up to 119 h post dose
Area under the concentration-time curve of S-bupropion in plasma over the time interval from 0 to the last quantifiable data point | up to 119 h post dose
Maximum measured concentration of total bupropion in plasma | up to 119 h post dose
Maximum measured concentration of S-bupropion in plasma | up to 119 h post dose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1307.20.1 Boehringer Ingelheim Investigational Site, Biberach, Germany